CLINICAL TRIAL: NCT07227922
Title: Clofutriben Pharmacokinetics in Patients With Impaired Renal Function
Acronym: RENAL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sparrow Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-62-CL-1005
Record Dates: First submitted 2025-11-06; First posted 2025-11-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Moderate Renal Impairment
Keywords: Renal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- clofutriben (Experimental)
  Interventions: Drug: 12mg clofutriben

INTERVENTIONS:
Drug: 12mg clofutriben — Each participant will receive a single oral dose of clofutriben

SUMMARY:
This is a Phase 1, single-center, open-label, single-dose trial. Sixteen participants are planned: 8 participants with moderate renal impairment and 8 matched control participants with normal renal function.

DETAILED DESCRIPTION:
Following Screening, enrolled participants will be confined to a clinical research unit for 6 days. Each participant will receive a single oral dose of clofutriben. Clofutriben PK, safety, and tolerability will be assessed. The participants will be contacted by telephone 4 weeks after clofutriben administration for safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants with stable moderate renal impairment (estimated glomerular filtration rate [eGFR]: 30 to <60 mL/min) and matched (by sex, age, and weight) control participants with normal renal function (eGFR: ≥90 mL/min) will be enrolled in this trial.

Exclusion Criteria:

* Participant whose current or recent medical conditions, medications, or procedures could increase participant's safety risk, or whom the Investigator considers not suitable for entry into the trial or the participant, or who has clinically significant abnormal 12-lead electrocardiogram (ECG)/ vital sign measurements/ laboratory test results at Screening and Check-in, will not be enrolled

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
1. Maximum plasma concentration (Cmax) | from enrollment through treatment for 6 days.
  Conclusions that clofutriben and AS2570469 exposures (separately) are not altered by moderate renal impairment will be reached if the 95% CIs of the geometric mean estimates of AUC0-t, AUC0-inf, and Cmax of clofutriben and AS2570469 fall within the [60%, 140%] range.
2. Area under the plasma time-concentration curve (AUC0-t, AUC0-inf) | from enrollment through treatment for 6 days.
  Conclusions that clofutriben and AS2570469 exposures (separately) are not altered by moderate renal impairment will be reached if the 95% CIs of the geometric mean estimates of AUC0-t, AUC0-inf, and Cmax of clofutriben and AS2570469 fall within the [60%, 140%] range.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States